CLINICAL TRIAL: NCT00416676
Title: UKCCSG Stage IIB/3 (INSS) Neuroblastoma Pilot Study [ENSG VI (Pilot 2B/3)]
Brief Title: Combination Chemotherapy and Surgery With or Without Radiation Therapy in Treating Patients With Stage 2 or Stage 3 Neuroblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-NB-1993-01; CDR0000454571 (Registry Identifier: PDQ (Physician Data Query)); EU-20594
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2006-12

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vincristine, cyclophosphamide, cisplatin, etoposide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving combination chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase III trial is studying how well giving combination chemotherapy and surgery with or without radiation therapy works in treating patients with stage 2 or stage 3 neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the acute and late toxicity of local radiotherapy when given after vincristine, cisplatin, etoposide, and cyclophosphamide (OPEC) alternating with vincristine, carboplatin, etoposide, and cyclophosphamide (OJEC) chemotherapy and surgery and followed by further chemotherapy in patients with stage 2B or 3 neuroblastoma.
* Determine the response in patients treated with alternating OPEC and OJEC chemotherapy before and after surgery.
* Determine the local control and event-free and overall survival of patients who achieve a complete response after chemotherapy and surgery alone.
* Determine the local control and event-free and overall survival of patients who do not achieve a complete response after chemotherapy and surgery and subsequently receive local radiotherapy.
* Determine clinical and biological prognostic factors for patients with stage 2B or 3 neuroblastoma when treated with this approach.

OUTLINE: This is a pilot, multicenter study.

Patients receive OPEC chemotherapy comprising vincristine IV and cyclophosphamide IV on day 1, cisplatin IV continuously over 24 hours on day 1, and etoposide IV over 4 hours on day 3 during courses 1, 3, and 5. Patients receive OJEC chemotherapy comprising vincristine IV, cyclophosphamide IV, etoposide IV over 4 hours, and carboplatin IV over 1 hour on day 1 during courses 2 and 4. Treatment repeats every 21 days for 5 courses. After 5 courses, patients with resectable disease undergo surgical resection. Patients who achieve a complete response (CR), either after surgery or after 5 courses of chemotherapy alone (where surgery is not possible), receive 2 additional courses of chemotherapy (OPEC followed by OJEC). Patients who do not achieve a CR undergo radiotherapy for 3 weeks. During the first week of radiotherapy, these patients also receive vincristine IV on day 1 and etoposide IV over 4 hours on days 1 and 2. Beginning 3 weeks after the completion of radiotherapy, these patients receive 2 additional courses of chemotherapy (OPEC followed by OJEC).

After completion of study treatment, patients are followed periodically for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma

  * Stage 2B or 3 disease
* Must be able to undergo radical radiotherapy

  * Radiotherapy contra-indicated if disease site is near a critical organ (e.g., mass overlying a single functioning kidney or the size of the residual tumor after chemotherapy precludes delivery of the specified radiation dose)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Barrett, Study Chair — University of Glasgow